CLINICAL TRIAL: NCT03143140
Title: The Clinical Value of Percutaneous Radiofrequency Ablation of Feeding Arterial for Hepatocellular Carcinoma
Brief Title: The Effect of Percutaneous Radiofrequency Ablation of Feeding Arterial for Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Kun Yan, Director of ultrasonography department, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Z151100004015186
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Liver Neoplasms
Keywords: Ablation Techniques
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAFA and tumor ablation (Experimental): first percutaneous frequency ablation of tumor feeding artery and then ablation of tumor
  Interventions: Other: PAFA; Other: tumor ablation
- tumor ablation (Other): ablation of tumor directly
  Interventions: Other: tumor ablation

INTERVENTIONS:
Other: PAFA — percutaneous ablation of tumor feeding artery
  Other Names: percutaneous ablation of tumor feeding artery
  Arms: PAFA and tumor ablation
Other: tumor ablation — ablation of tumor area directly

SUMMARY:
To evaluate a novel technique-ultrasound guided percutaneous abaltion of tumor feeding artery before RFA for liver malignancy.

DETAILED DESCRIPTION:
Hepatocellular carcinoma is one of the most common tumor in clinical practice. In recent years, various local therapies, especially radiofrequency ablation (RFA) has been proved safe and effective.The main limitation of RFA is that its therapeutic impact is significant compromised by blood flow cooling effect, especially in hypervascular HCC. Recent studies showed combined therapy of TACE and RFA can decrease the blood supply of tumor, increase ablated volume and therefore improve the outcome. However, TACE application is limited in patients who cannot tolerate this therapy due to the side effects of repeated TACE, poor liver function or previously legated hepatic artery. The present study is focus on "difficult-to-treat" HCC patients who are neither surgical candidates, nor TACE candidates. The investigators introduce the novel treatment mode that RFA followed ultrasound guided percutaneous ablation of tumur feeding arterial to treat these difficult cases and evaluate the clinical effect.

ELIGIBILITY:
Inclusion Criteria:

1. tumor number ≤3， maximum tumor size ≤5cm;
2. accessibility of tumors via a percutaneous approach;
3. tumor feeding artery can be detected by 3D contrast enhance ultrasound;
4. platelet count ≥ 50,000/ml and INR <1.6;
5. life expectancy more than 6 months
6. Child grade A or B

Exclusion Criteria:

1. patients who scheduled liver transplantation
2. with extrahepatic metastasis
3. women during menstruation, pregnancy, child birth and baby nursing period
4. patients with severe mental disorder
5. cardiopulmonary failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-05-22 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
completed tumor necrosis | 1 month
  Contrast enhanced CT or MRI was examed to evaluate tumor necrosis 1 month after ablation.

SECONDARY OUTCOMES:
tumor recurrence | up to 36 months
  tumor recurrence around the ablation zone

CONTACTS AND LOCATIONS:
Overall Officials: Kun Yan, master, Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang ZY, Lee JC, Yang W, Yan K, Wu W, Wang YJ, Chen MH. Percutaneous ablation of the tumor feeding artery for hypervascular hepatocellular carcinoma before tumor ablation. Int J Hyperthermia. 2018;35(1):133-139. doi: 10.1080/02656736.2018.1484525. Epub 2018 Jul 12. PMID 29999436